CLINICAL TRIAL: NCT00002931
Title: Tandem High-Dose Chemotherapy With Autologous Stem Cell Rescue for Poor-Prognosis Germ Cell Cancer
Brief Title: Combination Chemotherapy Plus Peripheral Stem Cell Transplantation in Treating Patients With Relapsed Germ Cell Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 96126; P30CA033572 (NIH); CHNMC-96126; NCI-G97-1136; CDR0000065365 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Results first posted 2017-01-04 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-01

CONDITIONS: Brain and Central Nervous System Tumors; Extragonadal Germ Cell Tumor; Ovarian Cancer; Teratoma; Testicular Germ Cell Tumor
Keywords: recurrent malignant testicular germ cell tumor; testicular seminoma; testicular embryonal carcinoma; testicular choriocarcinoma; testicular yolk sac tumor; testicular embryonal carcinoma and teratoma; testicular embryonal carcinoma and teratoma with seminoma; testicular embryonal carcinoma and yolk sac tumor; testicular embryonal carcinoma and yolk sac tumor with seminoma; testicular embryonal carcinoma and seminoma; testicular yolk sac tumor and teratoma; testicular yolk sac tumor and teratoma with seminoma; testicular choriocarcinoma and yolk sac tumor; testicular choriocarcinoma and embryonal carcinoma; testicular choriocarcinoma and teratoma; testicular choriocarcinoma and seminoma; recurrent ovarian germ cell tumor; recurrent extragonadal non-seminomatous germ cell tumor; recurrent extragonadal seminoma; recurrent extragonadal germ cell tumor; adult teratoma; testicular immature teratoma; testicular mature teratoma; ovarian immature teratoma; ovarian mature teratoma; ovarian monodermal and highly specialized teratoma; stage III malignant testicular germ cell tumor; stage IV ovarian germ cell tumor; stage IV extragonadal non-seminomatous germ cell tumor; stage IV extragonadal seminoma; adult central nervous system germ cell tumor
MeSH Terms: conditions — Central Nervous System Neoplasms; Ovarian Neoplasms; Teratoma; Testicular Germ Cell Tumor; Testicular Neoplasms; Seminoma; Endodermal Sinus Tumor; Carcinoma, Embryonal | interventions — Filgrastim; Carboplatin; Etoposide; Ifosfamide; Paclitaxel

ARMS (1):
- HD Chemo and Auto Stem Cells (Experimental)
  Interventions: Biological: filgrastim; Drug: carboplatin; Drug: etoposide; Drug: ifosfamide; Drug: paclitaxel; Procedure: autologous bone marrow transplantation; Procedure: bone marrow ablation with stem cell support

INTERVENTIONS:
Biological: filgrastim — 5 ug/kg bid beginning 4 days prior to and continuing through stem cell collection.
Drug: carboplatin — AUC=7, daily X 3
Drug: etoposide — 20 mg/kg by 2 hours infusion daily X 3
Drug: ifosfamide — 3 gm/m2 IV over 30 minutes X 3 days
Drug: paclitaxel — 425 mg/m2 as 24 hour continuous infusion
Procedure: autologous bone marrow transplantation — Given in two divided infusions on day -2 and day 0
Procedure: bone marrow ablation with stem cell support — Two cycles of high dose chemotherapy followed by stem cell reinfusion

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving combination chemotherapy together with bone marrow transplantation or peripheral stem cell transplantation works in treating patients with relapsed germ cell cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Estimate the antitumor activity of 2 courses of paclitaxel and carboplatin regimens with autologous stem cell rescue in patients with relapsed germ cell cancer.
* Evaluate the toxic effects of paclitaxel, carboplatin and etoposide (VP-16) with stem cell support followed by paclitaxel, carboplatin and ifosfamide with stem cell support in these patients.

OUTLINE: Patients receive filgrastim (G-CSF) SC or IV 4 days prior to peripheral blood stem cells (PBSC) apheresis. Autologous bone marrow harvest is performed when adequate stem cells cannot be collected.

Patients then receive course 1 of high-dose chemotherapy beginning on day -7 with paclitaxel IV over 24 hours. On days -6 to -4, patients receive etoposide IV over 2 hours and carboplatin (CBDCA) IV over 30 minutes 3 times daily. Following a 2 or 3 week recovery, a second course of chemotherapy begins on day -7, consisting of paclitaxel IV over 24 hours, then CBDCA and ifosfamide on days -6 to -4.

Reinfusion of PBSC and marrow begins on day -2 in both course 1 and 2. In addition, G-CSF IV is given twice a day until 3 consecutive postnadir days of granulocytes of at least 1000/mm^3 are maintained. On day 0, stem cells with or without bone marrow product are again administered.

Surgery may be performed after course 2 if indicated.

PROJECTED ACCRUAL: The expected accrual rate is 12 patients per year over 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Evaluable germ cell cancer (measurable by radiographic study and/or serum tumor marker elevation) and not curable by standard salvage therapy OR viable cancer on resection of post-chemotherapy residual masses in either intermediate or high risk category
* Bidimensionally measurable disease with measurements performed within 21 days of study entry
* Tumor marker (alpha-fetoprotein, lactate dehydrogenase, beta-human chorionic gonadotropin) studies performed within 7 days prior to study entry

PATIENT CHARACTERISTICS:

Age:

* 16 and over

Performance status:

* Karnofsky 70-100%

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 120,000/mm^3
* Hemoglobin at least 10 g/dL

Hepatic:

* Bilirubin no greater than 1.6 mg/dL
* SGOT and SGPT no greater than 2 times upper limit of normal (ULN)
* No active hepatitis or cirrhosis

Renal:

* Creatinine clearance at least 70 mL/min

Cardiovascular:

* Ejection fraction (MUGA or echocardiogram) normal
* No EKG evidence of active cardiac disease (arrhythmias, ischemia) which would contraindicate etoposide and paclitaxel study treatment

Pulmonary:

* PaO_2 at least 70 mm Hg
* FEV_1 at least 2 L or 75%
* No history of bleomycin associated or serious lung disease

Neurologic:

* No steroid or glucocorticoid treatment for patients with CNS metastatic disease; at least 1 month with stable post-radiotherapy neurological status and seizure free; if prior seizures, at least 1 month with therapeutic anticonvulsant levels prior to study
* Prior peripheral neuropathy requires consultation with principal investigator

Other:

* No significant active medical illness precluding study or survival
* Not HIV positive
* No prior malignancy within past 5 years except for adequately treated basal cell or squamous cell skin cancer
* No prior hematologic malignancies

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior bone marrow or stem cell rescue with high-dose chemotherapy

Chemotherapy:

* Prior chemotherapy allowed, excluding high-dose therapy with bone marrow or stem cell rescue
* No prior paclitaxel

Endocrine therapy:

* Not specified

Radiotherapy:

* No concurrent radiotherapy during study

Surgery:

* Recovered from prior surgery

Ages: 16 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 1997-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sumanta Pal, MD, Study Chair — City of Hope Medical Center
Locations (1):
- City of Hope Comprehensive Cancer Center, Duarte, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- HD Chemo and Auto Stem Cells: Cycle 1, stem cell mobilization with granulocyte-colony stimulating factor (G-CSF) at 10 μg/kg/d subcutaneously prior to leukapheresis. G-CSF administration daily during collection until the total collected product excelled 4 × 106 CD34+ cells/kg. 24-hour IV infusion of paclitaxel at 350 mg/m2 or 425 mg/m2 on day -7. Subsequent to this, patients receive etoposide (20 mg/kg IV over 2 hours) and carboplatin (AUC of 7 mg-min/mL IV over 30 minutes) daily on days -6, -5 and -4. IV infusion of 12.5% of the derived CD34+ stem cell product on day -2, followed by administration of 37.5% of the product on day 0. Cycle 2, comprised of paclitaxel, ifosfamide and carboplatin. Ifosfamide administered IV daily at 3 g/m2 over 30 minutes on days -6, -5 and -4. Mesna administered 24 hours subsequently as a 1 g/m2 bolus dose followed by 10g/m2 via continuous IV infusion over 72 hours. The derived CD34+ stem cell product administered in a manner identical to that during Cycle 1 on days -2 and 0.
Period: Overall Study
Arm/Group | HD Chemo and Auto Stem Cells
Started | 48
Completed | 46
Not Completed | 2
Not completed — rapidly progressing disease during | 2

BASELINE CHARACTERISTICS:
Arm/Group | HD Chemo and Auto Stem Cells
Number analyzed (Participants) | 48
Age, Continuous [Median (Full Range); unit: years] | 29 [16 to 49]
Gender [Count of Participants; unit: Participants]
  Female | 1
  Male | 47
Region of Enrollment [Number; unit: participants]
  United States | 48

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Estimated using the product-limit method of Kaplan and Meier. Progression is defined as an increase o any radiologically measureable tumor by greater than 25% or a greater than 10% increase of elevated tumor markers.
Time Frame: Until disease progression, up to 5 years.
Measure: Mean (95% Confidence Interval); unit: Months
Arm/Group | HD Chemo and Auto Stem Cells
Number analyzed (Participants) | 48
Months | 11.8 [5.8 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment.

2. Primary Outcome: Toxic Effects
Description: Number of Participants with Grade 3 and 4 Adverse Events Related to Protocol-based Therapy
Time Frame: From date of randomization until death of any cause, assessed up to 12 weeks
Measure: Number; unit: participants
Arm/Group | HD Chemo and Auto Stem Cells
Number analyzed (Participants) | 48
participants
  Hyperglycemia | 4
  Transaminase alone | 6
  Mucositis/stomatitis | 10
  Nausea/vomiting | 5
  Febrile neutropenia | 1
  Diarrhea | 3
  Hyperbilirubinemia | 3
  Fever w/o neutropenia | 2
  Hypocalcemia | 2
  Hemorrhage | 1
  Elevated INR/Prothrombin time | 2
  Renal Failure | 1
  Constipation | 1
  Esophagitis | 1

3. Secondary Outcome: Overall Survival
Description: Estimated using the product-limit method of Kaplan and Meier.
Time Frame: Until death from any cause, up to 5 years.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | HD Chemo and Auto Stem Cells
Number analyzed (Participants) | 48
Months | 21.7 [12.7 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment.

ADVERSE EVENTS:
Time Frame: Adverse events occurred over a period of 10 years and 6 months.
Description: "Other Adverse Events" include all events that were not severe adverse events regardless of grade or relation to treatment.
Arm/Group | HD Chemo and Auto Stem Cells
Serious Adverse Events (participants affected / at risk) | 1/48
Other Adverse Events (participants affected / at risk) | 46/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HD Chemo and Auto Stem Cells (N=48)
Renal failure (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HD Chemo and Auto Stem Cells (N=48)
Cerebellar (Nervous system disorders) | 15 (21)
Clinical (Physical Exam) (General disorders) | 13 (20)
Dysrhythmias (Cardiac disorders) | 9 (13)
Fluid Retention (General disorders) | 16 (25)
Hematemesis (Gastrointestinal disorders) | 3 (4)
Hemorrhage (Vascular disorders) | 16 (25)
Infection (Infections and infestations) | 16 (25)
Ischemia (Cardiac disorders) | 9 (13)
Other Misc (General disorders) | 14 (57)
Pericardial (Cardiac disorders) | 9 (13)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 16 (25)
Rash/desquamation associated with GVHD for BMT studies (Skin and subcutaneous tissue disorders) | 4 (5)
Stomatitis (Gastrointestinal disorders) | 16 (25)
Stomatitis/pharyngitis (oral/pharyngeal mucositis) for BMT studies, if specified in the protocol. (Gastrointestinal disorders) | 1 (1)
Weight (Food Intake) (Metabolism and nutrition disorders) | 7 (12)
Clinical Coagulation (Blood and lymphatic system disorders) | 10 (13)
Febrile neutropenia (ANC <1.0 x 10e9/L, fever >=38.5 degrees C) (Blood and lymphatic system disorders) | 12 (19)
Transfusion: Platelets (Blood and lymphatic system disorders) | 1 (1)
Transfusion: pRBCs (Blood and lymphatic system disorders) | 1 (1)
Cardiac ischemia/infarction (Cardiac disorders) | 1 (1)
EF/CHF (Cardiac disorders) | 9 (13)
Palpitations (Cardiac disorders) | 1 (1)
Supraventricular and nodal arrhythmia (Cardiac disorders) | 19 (25)
Auditory/Ear - Other (Specify, __) (Ear and labyrinth disorders) | 3 (6)
Hearing (Ear and labyrinth disorders) | 16 (21)
Cushingoid appearance (e.g., moon face, buffalo hump, centripetal obesity, cutaneous striae) (Endocrine disorders) | 1 (1)
Dry eye syndrome (Eye disorders) | 1 (1)
Ocular/Visual - Other (Specify, __) (Eye disorders) | 1 (4)
Ophthalmoplegia/diplopia (double vision) (Eye disorders) | 3 (3)
Vision (Eye disorders) | 16 (22)
Vision-blurred vision (Eye disorders) | 1 (1)
Watery eye (epiphora, tearing) (Eye disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 28 (39)
Diarrhea (Gastrointestinal disorders) | 41 (64)
Diarrhea patients with a colostomy (Gastrointestinal disorders) | 2 (4)
Esophagitis (Gastrointestinal disorders) | 2 (3)
Gastritis (including bile reflux gastritis) (Gastrointestinal disorders) | 1 (1)
Heartburn/dyspepsia (Gastrointestinal disorders) | 8 (9)
Incontinence (Gastrointestinal disorders) | 2 (2)
Melena/GI bleeding (Gastrointestinal disorders) | 3 (4)
Mucositis/stomatitis (functional/symptomatic) (Gastrointestinal disorders) | 29 (45)
Nausea (Gastrointestinal disorders) | 46 (74)
Proctitis (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 44 (73)
Edema (General disorders) | 15 (16)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1 (1)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 18 (26)
Fever (no infection) (General disorders) | 15 (22)
Injection site reaction/extravasation changes (General disorders) | 2 (2)
Pain - Other (Specify, __) (General disorders) | 11 (13)
Rigors/chills (General disorders) | 17 (25)
Hepatobiliary/Pancreas - Other (Specify, __) (Hepatobiliary disorders) | 2 (2)
Allergy (Immune system disorders) | 16 (25)
Infection (documented clinically or microbiologically) with ANC <1.0 x 10e9/L (Infections and infestations) | 1 (1)
Infection - Other (Specify, __) (Infections and infestations) | 1 (1)
Infection with unknown ANC (Infections and infestations) | 2 (2)
Infection without neutropenia (Infections and infestations) | 3 (4)
AGC (Investigations) | 16 (25)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 27 (42)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 27 (43)
Alkaline Phosphatase (Investigations) | 13 (20)
Alkaline phosphatase (Investigations) | 19 (24)
Amylase (Investigations) | 1 (1)
Bilirubin (Investigations) | 13 (20)
Bilirubin (hyperbilirubinemia) (Investigations) | 12 (15)
Creatinine (Investigations) | 26 (36)
HGB/HCT (Investigations) | 4 (5)
INR (International Normalized Ratio of prothrombin time) (Investigations) | 24 (38)
Neutrophils (ANC) (Somlo COH) (Investigations) | 7 (11)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 23 (39)
PTT (Partial Thromboplastin Time) (Investigations) | 16 (23)
Partial Thromboplastin Time (Investigations) | 10 (13)
Platelets (Investigations) | 38 (61)
Platelets (Somlo COH) (Investigations) | 7 (11)
Prothrombin Time (Investigations) | 10 (13)
SGOT/SGT (Investigations) | 13 (20)
WBC (Investigations) | 5 (7)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 3 (5)
Anorexia (Metabolism and nutrition disorders) | 13 (16)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 3 (3)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 29 (42)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 30 (46)
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 2 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 14 (21)
Hyperglycemia (Metabolism and nutrition disorders) | 15 (22)
Hypocalcemia (Metabolism and nutrition disorders) | 14 (21)
Hypoglycemia (Metabolism and nutrition disorders) | 15 (22)
Hypomagnesemia (Metabolism and nutrition disorders) | 15 (22)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 26 (39)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 2 (3)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 2 (2)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1 (2)
Cortical/State of Consciousness (Nervous system disorders) | 16 (22)
Dizziness (Nervous system disorders) | 8 (9)
Extrapyramidal/involuntary movement/restlessness (Nervous system disorders) | 4 (4)
Headache (Nervous system disorders) | 16 (22)
Motor Activity (Nervous system disorders) | 15 (21)
Neuropathy: motor (Nervous system disorders) | 19 (24)
Neuropathy: sensory (Nervous system disorders) | 25 (37)
Peripheral Nervous System Sensory (Nervous system disorders) | 15 (21)
Seizure (Nervous system disorders) | 1 (1)
Somnolence/depressed level of consciousness (Nervous system disorders) | 6 (6)
Speech impairment (e.g., dysphasia or aphasia) (Nervous system disorders) | 1 (1)
Syncope (fainting) (Nervous system disorders) | 1 (1)
Taste alteration (dysgeusia) (Nervous system disorders) | 5 (5)
Confusion (Psychiatric disorders) | 1 (1)
Hallucinations (Psychiatric disorders) | 3 (3)
Ideation (Psychiatric disorders) | 16 (22)
Insomnia (Psychiatric disorders) | 16 (21)
Mood (Psychiatric disorders) | 16 (22)
Mood alteration (Psychiatric disorders) | 18 (21)
Hematuria (Renal and urinary disorders) | 10 (15)
Hematuria (in the absence of vaginal bleeding) (Renal and urinary disorders) | 5 (6)
Pain (Renal and urinary disorders) | 22 (72)
Proteinuria (Renal and urinary disorders) | 11 (16)
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 1 (1)
Adult Respiratory Distress Syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hemorrhage, pulmonary/upper respiratory (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 11 (16)
Pulmonary/Upper Respiratory - Other (Specify, __) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Voice changes/dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dermatology/Skin - Other (Specify, __) (Skin and subcutaneous tissue disorders) | 10 (15)
Extensive Skin Rash (Skin and subcutaneous tissue disorders) | 13 (19)
Local Skin Rash (Skin and subcutaneous tissue disorders) | 13 (19)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 17 (24)
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 2 (2)
Acute vascular leak syndrome (Vascular disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (1)
Hemorrhage/Bleeding - Other (Specify, __) (Vascular disorders) | 9 (11)
Hypertension (Vascular disorders) | 13 (17)
Hypotension (Vascular disorders) | 19 (23)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes